CLINICAL TRIAL: NCT06661109
Title: Innovative Methods in Postsurgical Pain Management: A Randomized Controlled Trial on the Effects of Kinesio Taping After Cesarean Section
Brief Title: Innovative Methods in Postoperative Pain Management: A Study on the Effects of Kinesio Taping After Cesarean Section
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Collaborators: Toros University (Other)
Responsible Party: Principal Investigator, Yağmur SÜRMELİ, LECTURER DR., Toros University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TOROS UNIVERSITY
Record Dates: First submitted 2024-10-24; First posted 2024-10-28 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Over 18 Years Old
Keywords: kinesio-tape; kinesio-taping; comfort level; nurse; nursing
MeSH Terms: interventions — Methods; Population Groups

STUDY DESIGN:
Intervention Model Description: There will be 2 groups (intervention and placebo)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Taping (Experimental): Kinesio tape will be applied with 100% tension.
  Interventions: Other: Intervention (Kinesio Taping) group
- Sham Taping (Placebo Comparator): Kinesio tape will be applied without tension.
  Interventions: Other: Intervention (Kinesio Taping) group

INTERVENTIONS:
Other: Intervention (Kinesio Taping) group — No randomized study was found investigating the effect of kinesio taping on comfort levels in women having a cesarean delivery.

SUMMARY:
Brief Summary:

This randomized, single-blind study aimed to evaluate the effects of kinesio taping on pain management, comfort, and satisfaction of women after cesarean section.

The main question(s) it aimed to answer were:

* Is there a difference in mean pain scores between the intervention group and the control group as a result of kinesio taping?
* Is there a difference in mean comfort levels between the intervention group and the control group as a result of kinesio taping?

DETAILED DESCRIPTION:
The universe of this study will consist of women who underwent cesarean section surgery at the Gynecology and Obstetrics Clinic of a private hospital in the Mersin region between December 2024 and May 2025. The sample of the study will consist of women who meet the inclusion criteria and volunteer. The sample size was determined by the statistician using the G*Power 3.1.9.4 package program using a power analysis. The effect size (Cohen's d = 0.91) obtained based on the study conducted by Uzunkaya-Öztoprak (2019) and his colleagues was taken as the basis. At a power level of 90% and a significance level of 5%, a comparison of pain levels between the two groups (intervention and placebo) was planned and it was determined that at least 26 participants were required for each group. In order to prevent possible sample losses (20%), the sample size for each group was increased by 20% and therefore it was planned to include 31 participants in each group. Thus, it was anticipated that the study would be conducted with a total of 62 participants, and it was calculated that with this sample size, the study would have sufficient statistical power to meaningfully evaluate the effects on post-cesarean pain management, women's comfort and satisfaction.

Participants were assigned to the intervention and placebo groups using the randomization method in the study. The block randomization list used in assigning the groups will be made by an independent statistician other than the researchers using a random number table (https://www.randomizer.org/) to avoid bias. Data will be loaded into the program by assigning codes to the intervention and placebo groups and analyzed by an independent statistician instead of researchers who do not know the group codes. Thus, the study will also be blinded in terms of statistical analysis and reporting.Descriptive Characteristics Form, Visual Analog Scale, Perianesthesia Comfort Scale will be used to collect data.

Application Procedure Researcher Lecturer Yağmur Sürmeli (Y.S.) has received an internationally recognized "Kinesiology taping practitioner training certificate", which will make the implementation plan effective and efficient. Women who have cesarean delivery will be informed about the study in the clinic the day before the surgery (1 day before the surgery). Women who agree to participate in the study will sign the voluntary consent form. The inclusion and exclusion criteria of women who sign the informed consent form will be evaluated by the researchers. The study, which will be conducted by randomization, will consist of two groups: intervention (Kinesiology taping applied) and placebo (Sham taping applied). Before starting the kinesiology taping application, the "Information form on descriptive characteristics" and "Visual analog scale VAS" will be applied to the participants in both groups. All women in the study will be applied the routine nursing care and hospital analgesia protocol created for post-cesarean pain. Applications will be started 6-8 hours after the surgery due to the stabilization of the general condition and post-operative mobilization. During the applications, women's privacy will be protected and they will be asked not to remove the tapes until discharge. In addition, the tapes will be removed by the researcher at discharge.

Intervention Group: Taping will be applied to women in this group using 100% cotton, latex-free, 5 cm × 0.5 mm elastic tape Kinesio Tex GoldTM® (Kinesio Holding Corp., Albuquerque, NM, USA). If there is moisture such as sweat in the area where the taping will be applied that may affect the application, it will be wiped with a dry napkin. In order to increase the strength and support of the abdominal muscles after cesarean section, to provide muscle activation, to increase blood and lymph circulation and to reduce pain due to neurological suppression, two parallel and two vertical I tapes will be applied to the back and trochanter muscles with 100% tension as appropriate. Pain will be measured with VAS at the 1st hour after taping and at the 24th and 48th hours after surgery, and comfort will be evaluated with the "Perianesthesia Comfort Scale" before discharge.

Placebo Group: Women in this group will receive sham taping (tension-free kinesio taping). The quality of the kinesio taping used in the sham taping will be the same. Pain and comfort assessments will be made in the same way as in the intervention group.

Statistics Statistical analysis of the data will be performed using the IBM SPSS Statistics 24.0 (IBM SPSS Statistics for Windows, Version 24.0. Armonk, NY) program. Percentage, arithmetic mean and standard deviation will be calculated in the analysis of the data. In comparing the data between two groups, Independent Two Samples t-Test (if distribution is normal) or Mann-Whitney U Test (if distribution is not normal) will be performed for continuous variables, Chi-Square Test (if data is large enough) or Fisher's Exact Test (if sample is small) will be performed for categorical variables. Repeated Measures Analysis of Variance (ANOVA), if assumptions cannot be met, non-parametric tests such as Friedman Test will be used. Bonferroni correction will be applied for interactions. In all analyses, p<0.05 will be accepted as the statistical significance level.

Ethical Aspects of the Research Ethics committee and institutional approvals will be obtained for the study. The research will be conducted in accordance with the rules of the Declaration of Helsinki (World Medical Association, 2013). All women participating in the study will be informed and their written and verbal consent will be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-45
* Having undergone Caesarean section surgery and transverse incision technique
* Having undergone spinal or epidural anesthesia
* Having been classified as I or II by the American Society of Anesthesiologists (ASA)
* Having no dermatological, mental or perception problems
* Being open to communication
* Being willing to participate in the study

Exclusion Criteria:

* Having been diagnosed with an allergic skin disease,
* Developing postpartum complications (bleeding, infection, etc.),
* Expressing a desire to withdraw from the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women who have had a caesarean section
Enrollment: 62 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | At 1 hour after taping and at 24 and 48 hours postoperatively
  The Visual Analog Scale (VAS) is a method used to make some values that cannot be expressed numerically measurable. In this study, VAS will be used to determine the pain levels of women. Evaluation is made on a scale between 0 and 10 cm; 0 cm represents no pain, while 10 cm represents the most severe pain. On the scale, 0-44 mm is classified as mild pain, 45-74 mm as moderate pain, and 75-100 mm as severe pain. This test, which has been used for many years, is a widely accepted assessment tool known in the literature for its reliability and easy applicability.

SECONDARY OUTCOMES:
Perianesthesia Comfort Scale (PCS) | At 1 hour after taping and at 24 and 48 hours postoperatively
  The Perianesthesia Comfort Scale (PCS) determines the comfort levels of women who have had a cesarean delivery. The scale consists of 24 items and has a 6-point Likert-type scale. Statements range from "strongly disagree" to "strongly agree." Twelve of the items are positive (1, 5, 6, 11, 14, 16, 18, 19, 20, 21, 23, 24) and 12 are negative (2, 3, 4, 7, 8, 9, 10, 12, 13, 15, 17, 22), and the negative items are scored by reversing them. When evaluating the scale, the scores of the determined negative items are reverse-coded and added to the positive items. The highest total score that can be obtained from the scale is 144, and the lowest score is 24. The mean value is found by dividing the total scores by the number of items and the result is expressed as a distribution from 1 to 6. The Cronbach alpha coefficient of the scale is 0.89.

IPD SHARING:
Plan to Share IPD: No